CLINICAL TRIAL: NCT01517607
Title: Mesalazine (PENTASA®) in Ulcerative Colitis: Correlation of the Information Level With Patient's Compliance in Everyday Practice
Brief Title: Mesalazine (PENTASA®) in Ulcerative Colitis
Acronym: MUKOSA
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 000027
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mesalazine
  Interventions: Other: Mesalazine

INTERVENTIONS:
Other: Mesalazine — Patient's treated with oral Mesalazine

SUMMARY:
This non-interventional study examines whether the patient's level of information and the consideration of the patient's preference have a positive effect on the compliance and thus also on the therapeutic success.

ELIGIBILITY:
Inclusion Criteria:

* Patients are treated for the first time with oral PENTASA®, e.g. following first diagnosis of ulcerative colitis for treatment of an acute episode or
* Following a therapy-free period (no previous mesalazine therapy) or due to poor response or underdosage oder lacking acceptance of the previous medication the patients are re-adjusted to oral PENTASA®,
* The patients (≥ 18 years) have been informed about the NIS and have given their written consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care facilities
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patient compliance: Measured by patient response to a questionnaire | Month 0 - Month 12

SECONDARY OUTCOMES:
Patient's level of information: Measured by patient response to a questionnaire | Month 0 - Month 12
Patient's preference for the oral pharmaceutical form: Measured by patient response to a questionnaire | Month 0 - Month 12
Reasons for the therapeutic decision of the physician: Measured by physician responses | Month 0
Laboratory parameters of predefined blood measurements | Month 0- Month 12
  Faecal calprotectin (including test used), faecal lactoferrin. Number of leukocytes, C-reactive protein, blood sedimentation rate. Haemoglobin, serum iron, serum ferritin, transferrin saturation (TSAT)
Ulcerative Colitis Disease Activity Index (UCDAI) | Month 0 - Month 12
  UCDAI = Blood in stool, stool frequency, overall evaluation of the physician, endoscopic evaluation (optional)
Adverse drug reactions: measured by number of patients and event severity | Month 0 - Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (149):
- Germany (149):
  - Investigational site, Wettinerstraße 22, Altenburg
  - Investigational site, Marienstraße 6, Amberg
  - Investigational site, Adam-Ries-Straße 57c, Annaberg-Buchholz
  - Investigational site, Goethestraße 5, Ansbach
  - Investigational site, Elisenstraße 32, Aschaffenburg
  - Investigational site, Prinzregentenstraße 8, Augsburg
  - Investigational site, Koblenzer Straße 37, Bad Godesberg
  - Investigational site, Goethestraße 15g, Bad Neustadt an der Saale
  - Investigational site, Töpferstraße 17, Bautzen
  - Investigational site, Bahnhofstraße 18, Berlin
  - Investigational site, Blankenburger Chaussee 86, Berlin
  - Investigational site, Bundesallee 104-105, Berlin
  - Investigational site, Ehrenfelsstraße 47, Berlin
  - Investigational site, Etkar-Andre-Straße 8, Berlin
  - Investigational site, Hohenzollerndamm 47a, Berlin
  - Investigational site, Innsbrucker Straße 58, Berlin
  - Investigational site, Klosterstraße 34, Berlin
  - Investigational site, Kurfürstendamm 42, Berlin
  - Investigational site, Mohrenstraße 6, Berlin
  - Investigational site, Myslowitzer Straße 49, Berlin
  - Investigational site, Schönhauser Allee 118, Berlin
  - Investigational site, Schönhauser Allee 129, Berlin
  - Investigational site, Schönstraße 90, Berlin
  - Investigational site, Treskowallee 99, Berlin
  - Investigational site, Hauptstraße 88, Bielefeld
  - Investigational site, Hauptstraße 9, Bietigheim-Bissingen
  - Investigational site, Kasernenstraße 22-24, Bonn
  - Investigational site, Münsterstraße 18, Bonn
  - Investigational site, Propst-Sievert-Weg 9, Borken
  - Investigational site, Trauerberg 27-28, Brandenburg/Havel
  - Investigational site, Wetzlarer Straße 22, Butzbach
  - Investigational site, Hermann-Hesse-Platz 3, Calw
  - Investigational site, Dortmunder Straße, Castrop-Rauxl
  - Investigational site, Hainstraße 112, Chemnitz
  - Investigational site, Graseggerstraße 105, Cologne
  - Investigational site, Venloer Straße 247, Cologne
  - Investigational site, Bahnhofstraße 64, Cottbus
  - Investigational site, Vetschauer Straße 11a, Cottbus
  - Investigational site, Frankfurter Straße 3, Darmstadt
  - Investigational site, Rheinstraße 44-46, Darmstadt
  - Investigational site, Lagesche Straße 19, Detmold
  - Investigational site, Jahnstraße 1, Dingolfing
  - Investigational site, Karlsbader Straße 7, Dinkelsbühl
  - Investigational site, Recklinghäuser Straße 14, Dorsten
  - Investigational site, Rheinlanddamm 10, Dortmund
  - Investigational site, Lukasstraße 3, Dresden
  - Investigational site, Rehefelder Straße 12, Dresden
  - Investigational site, Mühlhäuser Straße 94, Haus F, Eisenach
  - Investigational site, Winkelgasse 1, Ellefeld
  - Investigational site, Königstraße 12-14, Elmshorn
  - Investigational site, Märkischestraße 30, Engelskirchen
  - Investigational site, Franz-Busbach-Straße 8, Erftstadt
  - Investigational site, Neuwerkstraße 2, Erfurt
  - Investigational site, Ruhrallee 81, Essen
  - Investigational site, Viktoriastraße 5, Euskirchen
  - Investigational site, Im Prüfling 23, Frankfurt
  - Investigational site, Hochstraße 43, Frankfurt am Main
  - Investigational site, Pfingsweidstraße 4, Frankfurt am Main
  - Investigational site, Stresemannallee 3, Frankfurt am Main
  - Investigational site, Habsburgerstraße 105, Freiburg im Breisgau
  - Investigational site, Schnetzenhauser Straße 5, Friedrichshafen
  - Investigational site, Moststraße 19, Fürth
  - Investigational site, Gartenstraße 29, Gardelegen
  - Investigational site, Hauptstraße 60-64, Garmisch-Partenkirchen
  - Investigational site, Am Markt 3, Gehrden
  - Investigational site, In der Heide 19, Gelsenkirchen
  - Investigational site, Von-der-Recke-Straße 14, Gelsenkirchen
  - Investigational site, Pollinger Straße 23, Gilching
  - Investigational site, Von-Werth-Straße 5, Grevenbroich
  - Investigational site, Avenwedder Straße 50, Gütersloh
  - Investigational site, Hachelweg 19, Hachelweg 19
  - Investigational site, Fürstin-Eugenie-Straße 7, Hachingen
  - Investigational site, Buscheystraße 15a, Hagen
  - Investigational site, Eppendorfer Baum 35-37, Hamburg
  - Investigational site, Eppendorfer Landstraße 42, Hamburg
  - Investigational site, Fontenay 1d, Hamburg
  - Investigational site, Harksheider Straße 3, Hamburg
  - Investigational site, Schlossstrasse 44, Hamburg
  - Investigational site, Schäferkampsallee 56-58, Hamburg
  - Investigational site, Sudetenweg 6, Hamm
  - Investigational site, Staufenbergstraße 31, Heilbronn
  - Investigational site, Frankfurter Straße 100a, Hennef (Sieg)
  - Investigational site, Am Ruschenhof 24, Herne
  - Investigational site, Wiescherstraße 20, Herne
  - Investigational site, Seestraße 43, Herrsching am Ammersee
  - Investigational site, Waisenhausstraße 2, Iserlohn
  - Investigational site, J.-Lange-straße 20, Jerichow
  - Investigational site, Prinzenallee 10, Jever
  - Investigational site, Hans-Sachs-Straße 1, Karlsruhe
  - Investigational site, Am Tiefen Weg 2, Karlstadt am Main
  - Investigational site, Opernstraße 9, Kassel
  - Investigational site, Feldstraße 5-7, Kiel
  - Investigational site, Moltkestraße 9, Kitzingen
  - Investigational site, Herzog-Adolph-Straße 13, Königstein
  - Investigational site, Schalaunische Straße 6-7, Köthen
  - Investigational site, Dreifaltigkeitsplatz 177, Landshut
  - Investigational site, Röntgenstraße 6-8, Langen
  - Investigational site, Funkenburgstraße 19, Leipzig
  - Investigational site, Johannisplatz 1, Leipzig
  - Investigational site, Markt 3, Leisnig
  - Investigational site, Am Gesundheitspark 11, Leverkusen
  - Investigational site, Yorckstraße 1, Ludwigshafen
  - Investigational site, Kronsforder Allee 19, Lübeck
  - Investigational site, Kronsforder Allee 69, Lübeck
  - Investigational site, Bismarckplatz 1, Mannheim
  - Investigational site, Stiftsweg 17, Mechernich
  - Investigational site, Am Harras 2, München
  - Investigational site, Irisstraße 23, München
  - Investigational site, Kaulbachstraße 61, München
  - Investigational site, Maximilianstraße 16, München
  - Investigational site, Schönfeldstraße 16, München
  - Investigational site, Unterer Markt 26-27, Neumarkt
  - Investigational site, Hofgründchen 13, Neuwied
  - Investigational site, Am Stadtpark 2, Nuremberg
  - Investigational site, Glogauer Straße 42, Nuremberg
  - Investigational site, Weiltinger Straße 11, Nuremberg
  - Investigational site, Hauptstraße 36, Oldenburg
  - Investigational site, Neue Donnerschweer Straße 30, Oldenburg
  - Investigational site, Ofener Straße 30, Oldenburg
  - Investigational site, Bramscher Straße 242, Osnabrück
  - Investigational site, Le-Mans-Wall 5, Paderborn
  - Investigational site, Westendstraße 38, Paderborn
  - Investigational site, Haptkanal rechts 75, Papenburg
  - Investigational site, Neundorfer Straße 14, Plauen
  - Investigational site, Allee nach Sanccouci 7, Potsdam
  - Investigational site, Großbeerenstraße 301, Potsdam
  - Investigational site, R.-Breitscheid-Straße 56, Potsdam
  - Investigational site, Kaiserstraße 166, Radevormwald
  - Investigational site, Neue Straße 34, Reinsdorf
  - Investigational site, Keramikerstraße 61, Rheinbach
  - Investigational site, St.-Petersburger-straße 18c, Rostock
  - Investigational site, Tegernseerstraße 100, Rottach-Weissach
  - Investigational site, Marktplatz 23, Rottenburg
  - Investigational site, Waldhausstraße 13, Schmalkalden
  - Investigational site, Krankenhausstraße 20, Schwalmstadt
  - Investigational site, Virchowstraße 10c, Singen
  - Investigational site, Wallstraße 38, Stade
  - Investigational site, Am Wallgraben 99, Stuttgart
  - Investigational site, Röhre 1, Sundern
  - Investigational site, Straße des Friedens 34c, Teuchern
  - Investigational site, Hambrocker Straße 53, Uelzen
  - Investigational site, Andreaestraße 16/1, Vahingen
  - Investigational site, Hochstraße 20, Waltrop
  - Investigational site, Kletzstraße 13B, Waren
  - Investigational site, Fischergasse 16, Weilheim
  - Investigational site, Julius-Leber-Strasße 8, Wesel
  - Investigational site, Westring 14, Wesseling
  - Investigational site, Forsthausstraße 1e, Wetzlar
  - Investigational site, Berliner Straße 8, Wittenberg